CLINICAL TRIAL: NCT01942447
Title: Fecal Microbiota Transplantation in Recurrent or Refractory Clostridium Difficile Colitis
Acronym: TOCSIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Martin Goetz, Univ.-Prof. Dr. med. Martin Goetz, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKT-FMT; UKT (Other: UKT)
Record Dates: First submitted 2013-09-05; First posted 2013-09-16 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Clostridium Difficile; Clostridium Difficile Infection
Keywords: Fecal microbiota transplantation; microbiota; clostridium difficile; clostridium difficile infection; Efficacy of FMT
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

ARMS (2):
- FMT (Experimental): FMT
  Interventions: Biological: FMT
- Standard (Active Comparator): Vancomycin
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Biological: FMT
  Arms: FMT
Drug: Vancomycin
  Arms: Standard

SUMMARY:
The host gastrointestinal microbiota is significantly influenced by antibiotic treatment which might favor Clostridium difficile infection (CDI), a frequent cause of community- and hospital-acquired, potentially life-threatening diarrhoea. CDI is followed by recurrence in 19-35% of patients despite adequate first line antimicrobial therapy. Currently there is no standardized therapy of recurrent or refractory CDI, but recent studies show remarkable effects of fecal microbiota transplantation (FMT).

In the current project, we aim to ideally match host and donor for FMT success in recurrent or refractory CDI. We will establish a clinical standard operating protocol for FMT, we will evaluate its safety and efficacy, and the patient acceptance and quality of life before and after FMT. We will analyse persistence of the donor microbiota within the recipient, define predictive clinical recipient and donor factors for FMT success and correlate them with microbial host and donor metagenomics.

We hypothesize that our work will yield novel, individualized strategies for recurrent or refractory CDI. In perspective, our results may be expanded to treatment of other inflammory bowel diseases.

ELIGIBILITY:
Inclusion Criteria:

* recurrent or refractory CDI
* previous antimicrobial therapy includes at least on course of vancomycin 4x125 (or higher doses) for at least 7d
* CDI, defined as: 3 or more loose bowel movements/d AND (presence of C.diff. toxin in stools or toxin producing C. diff. strain) OR (endoscopic or histologic evidence of pseudomembraneous colitis)

Exclusion Criteria:

* no informed consent
* no ability to provide informed consent
* immune suppression (continuous immune-suppressive drugs; steroids: prednisolone-equivalent > 20 mg for 14d or longer)
* lack of appropriate donor
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Resolution of diarrhea | 2 weeks
  Resolution of diarrhea

SECONDARY OUTCOMES:
Patient acceptance | 2 weeks

OTHER OUTCOMES:
Persitence of FMT | 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaetsklinikum Tuebingen, Tübingen, Germany